CLINICAL TRIAL: NCT00922012
Title: Efficacy of Electromagnetic Stimulation Therapy for the Treatment of Chronic Prostatitis or Chronic Pelvic Pain Syndrome
Brief Title: Efficacy of Electromagnetic Stimulation Therapy for Chronic Prostatitis and Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: M-cube technology (Unknown)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-08-064
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Prostatitis; Chronic Pelvic Pain Syndrome
Keywords: Electromagnetic Stimulation Therapy; Chronic Prostatitis; Chronic Pelvic Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electromagnetic stimulation (Experimental): Electromagnetic stimulation therapy
  Interventions: Device: Electromagnetic Stimulation Therapy

INTERVENTIONS:
Device: Electromagnetic Stimulation Therapy — Electromagnetic Stimulation Therapy for 24 weeks

SUMMARY:
In 1995 the National Institutes of Health-National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) workshop reached a consensus on the definition and classification of prostatitis syndromes.The commonest and yet most poorly understood of these prostatitis syndromes is category III or chronic pelvic pain syndrome (CPPS). It has been shown that, while men with CPPS have significantly higher leukocyte counts in urine and expressed prostatic secretions compared with age matched controls, inflammation and infection do not necessarily correlate with symptom severity.

The lack of a direct relationship between inflammation and symptoms is supported through studies of prostate histopathology, in which moderate or severe inflammation was identified in only 5% of men with CPPS.Conventional treatment has focused on long, empirical courses of expensive broad-spectrum antibiotics, mostly of the quinolone class, with or without the concomitant use of an α-blocker and anti-inflammatory agents. At the turn of the 19th century stimulation with electrical current and changing magnetic fields was used to treat surface conditions associated with intractable pain, such as painful malignant ulcers. The analgesic benefits of pulsed electromagnetic fields for relieving pelvic pain has been investigated in women with tissue trauma and chronic refractory pelvic pain.Despite its uncertain etiology there is some evidence that the symptom complex found in CPPS may be founded at least in part in pelvic floor muscular dysfunction and/or neurogenic hypersensitivity/inflammation.

We hypothesized that the application of a electromagnetic stimulation to the perineum of the subject may result in neural excitation and pelvic floor muscle stimulation to a degree that breaks the cycle of tonic muscular spasm and neural hypersensitivity/inflammation, thereby, restoring more normal pelvic floor muscular activity.

ELIGIBILITY:
Inclusion Criteria: male patients with

* Age ≥ 18
* NIDDK category III chronic prostatitis/chronic pelvic pain syndrome
* Symptom duration ≥ 3 months
* The sum of 1 or 2 domain of NIH-CPSI ≥ 1 point
* The sum NIH-CPSI ≥ 15 points

Exclusion Criteria: patients with

* History of prostate cancer
* History of pelvic irradiation
* History of transurethral surgery
* Urinary tract infection within 6 months to screening
* Postvoid urine volume ≥ 150ml
* Interstitial cystitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in NIH-CPSI total and pain score | 24 weeks after treatment

SECONDARY OUTCOMES:
Changes in - NIH-CPSI urinary, QoL impact score - Qmax/PVR - frequency/24hrs - urgency episode/24hrs - Patient perception of treatment benefit, satisfaction, willingness to continue - Goal achievement - Patient's Perception of Symptom Improvement | 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea